CLINICAL TRIAL: NCT05754346
Title: Does Inclusion of Diaphragmatic Breathing Exercises in Complete Decongestive Therapy Provide Further Benefits in Patients With Breast Cancer Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Bakircay University (Other)
Collaborators: Bezmialem Vakif University (Other); Istanbul Kent University (Other)
Responsible Party: Principal Investigator, Melih Zeren, asst. prof., Izmir Bakircay University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: bakircaymzeren07
Record Dates: First submitted 2023-02-22; First posted 2023-03-03 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Lymphedema, Breast Cancer; Lymphedema of Upper Limb
MeSH Terms: conditions — Breast Cancer Lymphedema

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (Active Comparator): Patients in this group will receive "Complete Decongestive Therapy" for 6 weeks. 1 session each week will be supervised in a clinic. Rest of the sessions will be performed at home.
  Interventions: Other: Complete Decongestive Therapy
- Study Group (Experimental): Patients in this group will receive "Complete Decongestive Therapy" combined with diaphragmatic breathing exercises for 6 weeks. 1 session each week will be supervised in a clinic. Rest of the sessions will be performed at home.
  Interventions: Other: Complete Decongestive Therapy; Other: Upper extremity exercises combined with diaphragmatic breathing exercises

INTERVENTIONS:
Other: Complete Decongestive Therapy — Complete Decongestive Therapy will include manual lymphedema drainage (self) for 20 min everyday, skin care everyday, wearing compression garment or bandages everyday and upper-extremity exercises twice a day.
Other: Upper extremity exercises combined with diaphragmatic breathing exercises — "Upper-extremity exercises" component of Complete Decongestive Therapy will be performed combined with diaphragmatic breathing exercises.
  Arms: Study Group

SUMMARY:
Complete decongestive therapy is proven to be effective in reducing lymphedema related symptoms such as swelling and pain. Breathing exercises, on the other hand, may also help managing lymphedema symptoms. Deep breathing creates a pressure change in the abdomen, which creates a vacuum effect in the thoracic cavity and helps to empty the lymphatic vessels. Thus, we aimed to investigate whether addition of diaphragmatic breathing exercises to physical exercise component of complete decongestive therapy provides further benefits on lymphedema volume, pain and quality of life in patients with breast cancer related lymphedema.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of arm lymphedema after being treated for unilateral breast cancer with axillary node dissection
* Completion of the treatments for the disease including chemotherapy and radiotherapy after breast surgery

Exclusion Criteria:

* Having recurrent cancer
* Having cognitive disability
* Having any concurrent diseases that may interfere with the measurement of lymphedema

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2023-03-20 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline lymphedema volume at 6th week | 6 weeks
  Arm volume will be measured using water displacement method.

SECONDARY OUTCOMES:
Change from baseline upper extremity pain at 6th week | 6 weeks
  Visual analog scale will be used for for quantifying pain.
Change from baseline quality of life at 6th week | 6 weeks
  Quality of life will be evaluated using Lymphedema Functioning, Disability and Health Questionnaire for Upper Limb Lymphedema.

CONTACTS AND LOCATIONS:
Overall Officials: Alis Kostanoglu, assoc.prof., Study Director — Bezmialem Vakif University
Locations (1):
- Bezmialem Vakif University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No